CLINICAL TRIAL: NCT04969783
Title: Telehealth Study Assessing the Removal of Filter Ventilation on Smoking Behavior and Biomarkers
Brief Title: Telehealth-Filter Ventilation ( COMET2P1 )
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021LS034; P01CA217806-S2 (Other Grant/Funding Number: NCI Trial ID); P01CA217806 (NIH)
Record Dates: First submitted 2021-07-06; First posted 2021-07-21 (Actual); Results first posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Tobacco Use
Keywords: cigarette smoking; filter ventilation
MeSH Terms: conditions — Tobacco Use; Cigarette Smoking

STUDY DESIGN:
Intervention Model Description: Phase III randomized, single blind, multi-center study assessing the impact of filter ventilation
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ventilated Cigarette Filter (Experimental): Filters with approximately 24-32% filter ventilation
  Interventions: Other: Ventilated Cigarette Filter
- Unventilated Cigarette Filter (Experimental): Filters with approximately 0-5.0% filter ventilation
  Interventions: Other: Unventilated Cigarette Filter

INTERVENTIONS:
Other: Ventilated Cigarette Filter — Ventilated Cigarette Filter
  Arms: Ventilated Cigarette Filter
Other: Unventilated Cigarette Filter — Unventilated Cigarette Filter
  Arms: Unventilated Cigarette Filter

SUMMARY:
The goals of this project are to determine the effects of varying degrees of cigarette filter ventilation on biomarkers of toxicant exposure and smoking behavior and on subjective responses to the cigarette.

The primary aim of this study is to examine the effects of unventilated vs ventilated filter cigarettes on urinary biomarkers of toxicant exposure and smoking behavior (e.g., cigarettes per day, intensity of smoking). The secondary objectives are 1) to examine the effects of cigarette filter ventilation on subjective measures such as cigarette dependence and responses to study cigarettes.

DETAILED DESCRIPTION:
This randomized controlled multi-site study will assess the effect of cigarettes with unventilated vs. ventilated filters on smoking behavior and biomarkers of tobacco toxicant exposure. The study, using telehealth and brief visits, will also examine the feasibility of remote collection of multiple biological samples.

Subjects (N=164; N=82 in each group) will be randomly assigned to: 1) Ventilated cigarettes; or 2) Unventilated cigarettes. Smokers will undergo an in person screening and then a 9 week experimental trial; 1 week of usual brand cigarettes; 2 weeks of ventilated study cigarettes and 6 weeks on either the ventilated or unventilated study cigarettes.

Subjective measures, alveolar carbon monoxide, blood pressure and cigarettes per day will be collected remotely. Biological samples collected at home will be dropped off at the clinic where the study cigarettes will be dispensed.

Biomarker samples will be assessed for total nicotine equivalents, tobacco specific nitrosamines and volatile organic compound.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age
* Biochemically confirmed regular cigarette smoker
* Daily smoker, 5-30 cigarettes per day.
* Usual brand cigarettes 16-36% ventilation

Exclusion Criteria:

* Unstable health
* Unstable medications
* Pregnant or nursing

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy K Hatsukami, Ph.D, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota Tobacco Research Program, Minneapolis, Minnesota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Intend to share findings from this research through publications and presentations. Institutions and individuals wishing to access any resources or data must contact the Principal Investigator (Hatsukami). Data will be available in two formats. One will be a summary of the data, with graphs and tables, posted as pdf files and as raw individual-level data for analysis. Data generated by this grant will be made to outside investigators, according to NIH Guidance. When data are shared, there will be no limits placed on how the data will be used. Users will agree, however, that the recipient must not transfer the data to other users and that the data are only to be used for research purposes. A record of transfer of data and a copy of the dataset that was distributed will be kept by University of Minnesota.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will not be available until primary and secondary papers are accepted for publication
Access Criteria: Persons requesting data must do so in writing, identifying their affiliation and how the data will be used. Upon review, access will be determined.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ventilated Cigarette Filter | Unventilated Cigarette Filter
Started | 80 | 84
Completed | 68 | 84
Not Completed | 12 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Physician Decision | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ventilated Cigarette Filter | Unventilated Cigarette Filter | Total
Number analyzed (Participants) | 80 | 84 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 78 | 83 | 161
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 48 | 100
  Male | 28 | 36 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 76 | 80 | 156
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 8 | 13
  White | 69 | 73 | 142
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 80 | 84 | 164

OUTCOME MEASURES:

1. Primary Outcome: Change in Total NNAL: 4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol [ng/g Creatinine]
Description: Absolute change from baseline level of total NNAL (4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol) at the week 6 visit (ng/g creatinine) measured in urine using liquid chromatography-tandem mass spectrometry (LC-MS/MS).
Time Frame: 6 weeks randomized intervention
Measure: Median (Inter-Quartile Range); unit: ng/g creatinine
Arm/Group | Ventilated Cigarette Filter | Unventilated Cigarette Filter
Number analyzed (Participants) | 67 | 82
ng/g creatinine | 0.97 [0.82 to 1.24] | 1.05 [0.84 to 1.35]

2. Primary Outcome: Change in Cigarettes Per Day (CPD)
Description: Change in cigarettes per day, daily diary reviewed data.
Time Frame: 7 days prior to week 0 visit and 7 days prior to week 6 visit
Measure: Mean (Standard Deviation); unit: Cigarettes per day
Arm/Group | Ventilated Cigarette Filter | Unventilated Cigarette Filter
Number analyzed (Participants) | 68 | 84
Cigarettes per day | -0.39 (2.73) | -0.17 (3.41)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Ventilated Cigarette Filter | Unventilated Cigarette Filter
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/84
Serious Adverse Events (participants affected / at risk) | 1/80 | 0/84
Other Adverse Events (participants affected / at risk) | 73/80 | 74/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ventilated Cigarette Filter (N=80) | Unventilated Cigarette Filter (N=84)
Superficial blood clot in lower leg (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ventilated Cigarette Filter (N=80) | Unventilated Cigarette Filter (N=84)
Nasal congestion (incl. runny nose) (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 8 (9)
Headache (incl. migraine) (Nervous system disorders) | 7 (8) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (10)
Sore/itchy/irritated throat (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (10)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2)
COVID-19 (Infections and infestations) | 3 (3) | 4 (4)
Fatigue (General disorders) | 3 (3) | 4 (4)
Myalgia (muscle aches/pain/spasms) (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Cough, Productive (lung 'fullness') (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Allergic rhinitis (incl. seasonal allergies) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Depressed (sad) mood (Psychiatric disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1)
Hypertension / Elevated BP (Vascular disorders) | 2 (2) | 2 (2)
Pain (other) (General disorders) | 1 (1) | 0 (0)
Anxious (nervous) mood (Psychiatric disorders) | 0 (0) | 3 (3)
Fever (General disorders) | 2 (2) | 1 (1)
Ear Pain (ache/fullness) (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Chills (General disorders) | 2 (2) | 1 (1)
Infections and Infestations - Other, Specify (Infections and infestations) | 2 (2) | 1 (1)
Tachycardia / Fast heart rate (Cardiac disorders) | 1 (1) | 1 (1)
Oral dysesthesia (burning/tingling/numbness/pain) (Gastrointestinal disorders) | 1 (1) | 1 (1)
Sinus Pain (Nervous system disorders) | 0 (0) | 1 (1)
Surgical and medical procedures, Other, Specify (Surgical and medical procedures) | 1 (1) | 0 (0)
Dysgeusia (change in taste/smell) (Nervous system disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Influenza (PCP dx; cough/lung sx separately) (Infections and infestations) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sinusitis - sinus infection (incl. bacterial, fungal, viral) (Infections and infestations) | 1 (1) | 0 (0)
Neuralgia / Neuropathy (nerve pain) (Nervous system disorders) | 0 (0) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Investigations - Other abnormal lab, low blood oxygen (Investigations) | 1 (1) | 0 (0)
Gastroesophageal Reflux (GERD/heartburn/acid) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypotension / Low BP (Vascular disorders) | 1 (1) | 0 (0)
Sprained joint (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Phlegm, increase in (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/83/NCT04969783/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT04969783/ICF_001.pdf